CLINICAL TRIAL: NCT00446797
Title: An Open Label Randomized Multicenter Comparative Study On Celecoxib Efficacy And Safety Versus Non-Selective NSAID In Acute Pain Due To Ankle Sprain
Brief Title: Open Label Comparative Study On Celecoxib Efficacy And Safety Vs Non-Selective NSAID In Acute Pain Due To Ankle Sprain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A3191332
Record Dates: First submitted 2007-03-09; First posted 2007-03-13 (Estimated); Results first posted 2009-06-10 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Ankle Sprain
Keywords: Ankle sprain, acute pain, NSAID, celecoxib,
MeSH Terms: conditions — Ankle Injuries; Acute Pain | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-Selective NSAIDS (Active Comparator): nsNSAIDs used in real-life standard practice for treatment of pain due to ankle sprain.
  Interventions: Drug: Non-selective NSAIDS
- Celecoxib (Experimental)
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Non-selective NSAIDS — Non-selective NSAIDs administered at usual (standard) doses.
  Arms: Non-Selective NSAIDS
Drug: Celecoxib — celecoxib with an initial loading dose of 400 mg followed by 200 mg twice daily (BID) for up to 7 days.
  Arms: Celecoxib

SUMMARY:
To assess the efficacy of celecoxib loading dose of 400mg followed by 200 mg twice a day (BID) versus oral non-selective NSAIDs in acute pain due to ankle sprain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with first acute ankle sprain episode in the last six months classified as grade I or II, confirmed by X-rays, according to the following definitions:
* Grade I: When the ligament is stretched but not torn and the anterior talofibular ligament is usually involved. The anterior draw test is negative.
* Grade II: Moderate sprains which usually result in partial tears af the ligaments, primarily the anterior talofibular and possibly the calcaneofibular ligament. Ligamentous laxity may be present and there is moderate swelling.

Exclusion Criteria:

* Patients who have a similar injury of the same joint within the last six months; or
* clinical evidence of complete rupture of ankle ligaments (third degree sprain), or
* requirements for bed rest, hospitalization, surgical intervention for the ankle injury; or
* evidence of fractures; or non-removable full cast of any tipe; or
* presence of bilateral occurrence of ankle injury or ipsilateral ankle and knee injury.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2007-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- Brazil (3):
  - Pfizer Investigational Site, Goiânia, Goiás
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, São Paulo, São Paulo
- Pfizer Investigational Site, San Antonio Guadalupe, Guadalupe, San Jose, Costa Rica
- Pfizer Investigational Site, Quito, Pichincha, Ecuador
- Pfizer Investigational Site, Cairo, Egypt
- Pfizer Investigational Site, Amman, Jordan
- Mexico (4):
  - Pfizer Investigational Site, Mexico City, Mexico City
  - Pfizer Investigational Site, San Nicolás de los Garza, Nuevo León
  - Pfizer Investigational Site, Toluca, State of Mexico
  - Pfizer Investigational Site, México DF
- Pfizer Investigational Site, Panama City, Panama
- Pfizer Investigational Site, Lima, Peru

REFERENCES:
- [Derived] Jones P, Lamdin R, Dalziel SR. Oral non-steroidal anti-inflammatory drugs versus other oral analgesic agents for acute soft tissue injury. Cochrane Database Syst Rev. 2020 Aug 12;8(8):CD007789. doi: 10.1002/14651858.CD007789.pub3. PMID 32797734
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191332&StudyName=Open%20Label%20Comparative%20Study%20On%20Celecoxib%20Efficacy%20And%20Safety%20Vs%20Non-Selective%20NSAID%20In%20Acute%20Pain%20Due%20To%20Ankle%20Sprain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Locations used were emergency rooms at orthopedic hospitals, general hospitals or private doctor's offices
Pre-assignment Details: Subjects sustained ankle sprain with a pain rating of greater than or equal to 45mm on a visual analog scale on full weight bearing, no more than 48 hours prior to the first dose of study medication
Groups:
- Celecoxib: All participants randomized to celecoxib were treated with 2 capsules of celecoxib 200 mg as a loading dose, thereafter, participants took 1 capsule of celecoxib 200 mg twice daily (morning and evening), for up to 7 days. Approximately a 12 hour interval was maintained between doses.
- nsNSAIDs: All participants randomized to non-selective non-steroidal anti inflammatory drugs (nsNSAIDs) took the first dose and all subsequent doses according to the standard treatment practice for treatment of pain due to ankle sprain, for up to 7 days.
Period: Overall Study
Arm/Group | Celecoxib | nsNSAIDs
Started | 141 | 137
Completed | 133 | 125
Not Completed | 8 | 12
Not completed — Lack of Efficacy | 0 | 2
Not completed — Lost to Follow-up | 5 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Protocol Violation | 1 | 3
Not completed — subject entered at another site | 0 | 1
Not completed — did not meet entrance criteria | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Celecoxib | nsNSAIDs | Total
Number analyzed (Participants) | 141 | 137 | 278
Age, Continuous [Mean (Full Range); unit: years] | 30.6 [18 to 66] | 30.4 [18 to 74] | 30.5 [18 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 55 | 111
  Male | 85 | 82 | 167

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Day 3 in Pain Visual Analog Scale (VAS) - Per Protocol Population
Description: Assessment of ankle pain by VAS: 100 mm horizontal line with left end being "No Pain" & right end being "Worst Possible Pain". Participants drew vertical line on horizontal scale to best reflect current pain on full weight bearing of injured ankle. Distance from left end of line to mark. Change: mean score at day 3 minus mean score at baseline
Time Frame: Baseline and day 3
Population: Per protocol (PP) population included subjects who were randomized, received full loading dose of study medication on day 1 and took no prohibited medications up to and including day 3, had valid baseline and day 3 VAS scores and had no major protocol violations before or during the study (i.e. a subset of treated subjects).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 131 | 126
scores on a scale | -44.88 (19.75) | -40.76 (18.91)
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Least squares mean; Test type: Non-Inferiority or Equivalence — To conclude non inferiority, the lower bound of the 2-sided 95% confidence interval of the difference in change scores between the 2 treatment groups (nsNSAIDs - celecoxib) must be greater than -10 mm; ANCOVA; Terms for treatment, country (fixed), and the baseline pain VAS score; Mean Difference (Final Values) = 3.39, 95% CI [-0.76 to 7.55], Standard Error of Mean 2.11 — Direction: nsNSAIDs minus celecoxib

2. Secondary Outcome: Change From Baseline in Pain Visual Analog Scale (VAS) - Modified Intent to Treat Population
Description: Assessment of ankle pain by VAS: 100 mm horizontal line, left end being "No Pain" & right end being "Worst Possible Pain". Participants drew vertical line on horizontal scale to best reflect current pain on full weight bearing of injured ankle. Distance from left end of line to mark. Change: mean score at observation minus mean score at baseline
Time Frame: Baseline and days 2, 3 and 7
Population: Modified intent to treat (MITT) population included subjects who were randomized, received at least one dose of study medication and had at least one follow up pain VAS score assessment (i.e. a subset of treated subjects).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 135 | 133
scores on a scale
  Day 2 | -29.25 (18.99) | -25.98 (18.21)
  Day 3 | -44.87 (19.51) | -40.75 (18.74)
  Day 7 | -61.17 (18.43) | -57.89 (18.84)
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Day 2 Least squares mean; Test type: Superiority or Other; ANCOVA; Terms for treatment, country (fixed) and the baseline pain VAS score; Mean Difference (Final Values) = 3.10, 95% CI [-0.89 to 7.08], Standard Error of Mean 2.02 — Direction: nsNSAIDs minus celecoxib
Statistical Analysis 2: Comparison: Celecoxib vs nsNSAIDs; Day 3 Least squares mean; Test type: Superiority or Other; ANCOVA; Terms for treatment, country (fixed) and the baseline pain VAS score; Mean Difference (Final Values) = 3.46, 95% CI [-0.55 to 7.48], Standard Error of Mean 2.04 — Direction: nsNSAIDs minus celecoxib
Statistical Analysis 3: Comparison: Celecoxib vs nsNSAIDs; Day 7 Least squares mean; Test type: Superiority or Other; ANCOVA; Terms for treatment, country (fixed) and the baseline pain VAS score; Mean Difference (Final Values) = 2.76, 95% CI [-0.91 to 6.42], Standard Error of Mean 1.86 — Direction: nsNSAIDs minus celecoxib

3. Secondary Outcome: Number of Subjects Responding (Improving) - MITT Population
Description: The number of subjects showing a response: a decrease of at least 20 mm (that is improvement) on the pain visual analog scale (VAS) scale
Time Frame: Days 2, 3 and 7
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 135 | 133
participants
  Day 2 - response (N=134, 133) | 91 | 79
  Day 2 - no response | 43 | 54
  Day 3 - response (N=135, 131) | 124 | 116
  Day 3 - no response | 11 | 15
  Day 7 - response (N=133, 125) | 129 | 120
  Day 7 - no response | 4 | 5
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Day 2; Test type: Superiority or Other; p = 0.1591, Regression, Logistic — Threshold for statistical significance: p value is less than or equal to 0.05; Terms for treatment and the baseline pain VAS score
Statistical Analysis 2: Comparison: Celecoxib vs nsNSAIDs; Day 3; Test type: Superiority or Other; p = 0.3995, Regression, Logistic — Threshold for statistical significance: p value is less than or equal to 0.05; Terms for treatment and the baseline pain VAS score
Statistical Analysis 3: Comparison: Celecoxib vs nsNSAIDs; Day 7; Test type: Superiority or Other; p = 0.6805, Regression, Logistic — Threshold for statistical significance: p value is less than or equal to 0.05; Terms for treatment and the baseline pain VAS score

4. Secondary Outcome: Subject's Global Assessment of Ankle Injury
Description: Subject response to question: "Considering all the ways your ankle injury affects you, how are you doing today?" Scale: 5 point from 1 = very good (no symptoms and no limitation of normal activities) to 5 = very poor (very severe symptoms which are intolerable and inability to carry out all normal activities).
Time Frame: Days 2, 3 and 7
Population: Modified intent to treat (MITT) population included subjects who were randomized, received at least one dose of study medication and had at least one follow up pain VAS score assessment
Measure: Number; unit: participants
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 135 | 133
participants
  Day 2 - Very good (no symptoms) (N=135, 133) | 1 | 1
  Day 2 - Good (mild symptoms) | 40 | 31
  Day 2 - Fair (moderate symptoms) | 76 | 80
  Day 2 - Poor (severe symptoms) | 17 | 19
  Day 2- Very poor (very severe symptoms) | 1 | 2
  Day 3 - Very good (no symptoms) (N=135, 131) | 8 | 6
  Day 3 - Good (mild symptoms) | 68 | 55
  Day 3 - Fair (moderate symptoms) | 54 | 63
  Day 3 - Poor (severe symptoms) | 5 | 7
  Day 3 - Very poor (very severe symptoms) | 0 | 0
  Day 7 - Very good (no symptoms) (N=133, 125) | 53 | 37
  Day 7 - Good (mild symptoms) | 61 | 63
  Day 7 - Fair (moderate symptoms) | 17 | 21
  Day 7 - Poor (severe symptoms) | 2 | 4
  Day 7 - Very poor (very severe symptoms) | 0 | 0
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Day 2; Test type: Superiority or Other; p = 0.2411, Cochran-Mantel-Haenszel — Threshold for statistical significance: p value is less than or equal to 0.05; Controlled for country Test of row mean score differences based on modified ridits (standardizing the mid-rank)
Statistical Analysis 2: Comparison: Celecoxib vs nsNSAIDs; Day 3; Test type: Superiority or Other; p = 0.1163, Cochran-Mantel-Haenszel — Threshold for statistical significance: p value is less than or equal to 0.05; Controlled for country Test of row mean score differences based on modified ridits (standardizing the mid-rank)
Statistical Analysis 3: Comparison: Celecoxib vs nsNSAIDs; Day 7; Test type: Superiority or Other; p = 0.0440, Cochran-Mantel-Haenszel — Threshold for statistical significance: p value is less than or equal to 0.05; Controlled for country Test of row mean score differences based on modified ridits (standardizing the mid-rank)

5. Secondary Outcome: Physician Global Assessment of Ankle Injury
Description: Investigator evaluation of overall severity of ankle injury. Scale: 5 point from 1 = Very mild (very mild signs and symptoms of ankle sprain) to 5 =Very severe (very severe signs and symptoms of ankle sprain)
Time Frame: Days 3 and 7
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 135 | 133
participants
  Day 3 - very mild (N=134, 131) | 20 | 12
  Day 3 - mild | 71 | 79
  Day 3 - moderate | 40 | 38
  Day 3 - severe | 2 | 2
  Day 3 - very severe | 1 | 0
  Day 7 - very mild (N=132, 125) | 87 | 70
  Day 7 - mild | 38 | 47
  Day 7 - moderate | 7 | 7
  Day 7 - severe | 0 | 1
  Day 7 - very severe | 0 | 0
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Day 3; Test type: Superiority or Other; p = 0.7223, Cochran-Mantel-Haenszel — Threshold for statistical significance: p value is less than or equal to 0.05; Controlled for country Test of row mean score differences based on modified ridits (standardizing the mid-rank)
Statistical Analysis 2: Comparison: Celecoxib vs nsNSAIDs; Day 7; Test type: Superiority or Other; p = 0.0541, Cochran-Mantel-Haenszel — Threshold for statistical significance: p value is less than or equal to 0.05; Controlled for country Test of row mean score differences based on modified ridits (standardizing the mid-rank)

6. Secondary Outcome: Pain Relief - MITT Population
Description: Subject's response to the statement "My relief from starting pain is". Scale from 0 = None to 4 = Complete.
Time Frame: Days 2, 3 and 7
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 135 | 133
participants
  Day 2 - None (N=135, 132) | 8 | 5
  Day 2 - A little | 25 | 33
  Day 2 - Some | 49 | 52
  Day 2 - A lot | 52 | 42
  Day 2 -Complete | 1 | 0
  Day 3 - None (N=135, 131) | 0 | 1
  Day 3 - A little | 15 | 21
  Day 3 - Some | 33 | 46
  Day 3 - A lot | 84 | 60
  Day 3 -Complete | 3 | 3
  Day 7 - None (N=133, 125) | 1 | 1
  Day 7 - A little | 6 | 3
  Day 7 - Some | 7 | 15
  Day 7 - A lot | 77 | 80
  Day 7 -Complete | 42 | 26
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Day 2; Test type: Superiority or Other; p = 0.2900, Cochran-Mantel-Haenszel — Threshold for statistical significance: p value is less than or equal to 0.05; Controlled for country Test of row mean score differences based on modified ridits (standardizing the mid-rank)
Statistical Analysis 2: Comparison: Celecoxib vs nsNSAIDs; Day 3; Test type: Superiority or Other; p = 0.0157, Cochran-Mantel-Haenszel — Threshold for statistical significance: p value is less than or equal to 0.05; Controlled for country Test of row mean score differences based on modified ridits (standardizing the mid-rank)
Statistical Analysis 3: Comparison: Celecoxib vs nsNSAIDs; Day 7; Test type: Superiority or Other; p = 0.1206, Cochran-Mantel-Haenszel — Threshold for statistical significance: p value is less than or equal to 0.05; Controlled for country Test of row mean score differences based on modified ridits (standardizing the mid-rank)

7. Secondary Outcome: Subject Assessment of Normal Function / Activity
Description: Subject response to question: "How does your ankle injury affect your walking and normal activity?" Scale from 1 = Normal walking/activity and no pain to 5 = Severely restricted walking due to pain and can't resume normal activities (normal activities defined as all activity that a subject did on a routine basis, including work and recreation)
Time Frame: Days 2, 3 and 7
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 135 | 133
participants
  Day 2 - normal no pain (N =135, 133) | 5 | 2
  Day 2 - normal with pain | 40 | 30
  Day 2 - mildly restricted | 59 | 55
  Day 2 - moderately restricted | 19 | 39
  Day 2 - severely restricted | 12 | 7
  Day 3 - normal no pain (N = 135, 131) | 18 | 13
  Day 3 - normal with pain | 52 | 46
  Day 3 - mildly restricted | 49 | 57
  Day 3 - moderately restricted | 14 | 11
  Day 3 - severely restricted | 2 | 4
  Day 7 - normal no pain (N = 133, 125) | 62 | 43
  Day 7 - normal with pain | 55 | 68
  Day 7 - mildly restricted | 11 | 8
  Day 7 - moderately restricted | 4 | 3
  Day 7 - severely restricted | 1 | 3
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Day 2; Test type: Superiority or Other; p = 0.0846, Cochran-Mantel-Haenszel — Threshold for statistical significance: p value is less than or equal to 0.05; Controlled for country Test of row mean score differences based on modified ridits (standardizing the mid-rank)
Statistical Analysis 2: Comparison: Celecoxib vs nsNSAIDs; Day 3; Test type: Superiority or Other; p = 0.3041, Cochran-Mantel-Haenszel — Threshold for statistical significance: p value is less than or equal to 0.05; Controlled for country Test of row mean score differences based on modified ridits (standardizing the mid-rank)
Statistical Analysis 3: Comparison: Celecoxib vs nsNSAIDs; Day 7; Test type: Superiority or Other; p = 0.1216, Cochran-Mantel-Haenszel — Threshold for statistical significance: p value is less than or equal to 0.05; Controlled for country Test of row mean score differences based on modified ridits (standardizing the mid-rank)

8. Secondary Outcome: Modified Brief Pain Inventory Short Form (m-BPI-sf) - Pain Severity Question 1
Description: m-BPI-sf questionnaire assessed pain severity and pain interference with functional activities during the 24 hour follow-up period.
  Q1: Subject response to 'describe your pain at its worst in the last 24 hours'. Scale: 0 = no pain to 10 = pain as bad as you can imagine
Time Frame: Days 1, 3 and 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 135 | 133
scores on a scale
  Day 2 (N = 134, 133) | 5.71 (2.04) | 5.90 (2.06)
  Day 3 (N = 135, 131) | 3.81 (1.84) | 4.44 (1.91)
  Day 7 (N = 133, 125) | 2.08 (1.93) | 2.38 (1.78)
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Day 2 Least squares mean; Test type: Superiority or Other; p = 0.395, ANCOVA — Overall p-value; Terms for treatment and country; Mean Difference (Final Values) = 0.14, 95% CI [-0.33 to 0.62], Standard Error of Mean 0.24 — Direction: nsNSAIDs minus celecoxib
Statistical Analysis 2: Comparison: Celecoxib vs nsNSAIDs; Day 3 Least squares mean; Test type: Superiority or Other; p = 0.004, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = 0.61, 95% CI [0.18 to 1.04], Standard Error of Mean 0.22 — Direction: nsNSAIDs minus celecoxib
Statistical Analysis 3: Comparison: Celecoxib vs nsNSAIDs; Day 7 Least squares mean; Test type: Superiority or Other; p = 0.122, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = 0.35, 95% CI [-0.08 to 0.77], Standard Error of Mean 0.22 — Direction: nsNSAIDs minus celecoxib

9. Secondary Outcome: Modified Brief Pain Inventory Short Form (m-BPI-sf) - Pain Severity Question 2
Description: m-BPI-sf questionnaire assessed pain severity and pain interference with functional activities during the 24 hour follow-up period.
  Q2: Subject response to 'describe your pain at its least in the last 24 hours'. Scale: 0 = no pain to 10 = pain as bad as you can imagine
Time Frame: Days 2, 3 and 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 135 | 133
scores on a scale
  Day 2 (N = 133, 133) | 3.25 (1.83) | 3.36 (1.88)
  Day 3 (N = 135, 131) | 2.07 (1.68) | 2.40 (1.64)
  Day 7 (N = 133, 125) | 0.83 (1.26) | 1.16 (1.43)
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Day 2 Least squares mean; Test type: Superiority or Other; p = 0.604, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = 0.09, 95% CI [-0.32 to 0.49], Standard Error of Mean 0.21 — Direction: nsNSAIDs minus celecoxib
Statistical Analysis 2: Comparison: Celecoxib vs nsNSAIDs; Day 3 Least squares mean; Test type: Superiority or Other; p = 0.124, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = 0.28, 95% CI [-0.07 to 0.63], Standard Deviation 0.18 — Direction: nsNSAIDs minus celecoxib
Statistical Analysis 3: Comparison: Celecoxib vs nsNSAIDs; Day 7 Least squares mean; Test type: Superiority or Other; p = 0.062, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = 0.32, 95% CI [0.03 to 0.61], Standard Error of Mean 0.15 — Direction: nsNSAIDs minus celecoxib

10. Secondary Outcome: Modified Brief Pain Inventory Short Form (m-BPI-sf) - Pain Severity Question 3
Description: m-BPI-sf questionnaire assessed pain severity and pain interference with functional activities during the 24 hour follow-up period.
  Q3: Subject response to 'describe your pain on the average'. Scale: 0 = no pain to 10 = pain as bad as you can imagine
Time Frame: Days 2, 3 and 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 135 | 133
scores on a scale
  Day 2 (N = 134, 133) | 4.34 (1.79) | 4.41 (1.90)
  Day 3 (N = 135, 131) | 2.90 (1.70) | 3.26 (1.63)
  Day 7 (N = 133, 125) | 1.41 (1.56) | 1.74 (1.53)
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Day 2 Least squares mean; Test type: Superiority or Other; p = 0.705, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = 0.05, 95% CI [-0.36 to 0.47], Standard Error of Mean 0.21 — Direction: nsNSAIDs minus celecoxib
Statistical Analysis 2: Comparison: Celecoxib vs nsNSAIDs; Day 3 Least squares mean; Test type: Superiority or Other; p = 0.064, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = 0.36, 95% CI [-0.01 to 0.73], Standard Error of Mean 0.19 — Direction: nsNSAIDs minus celecoxib
Statistical Analysis 3: Comparison: Celecoxib vs nsNSAIDs; Day 7 Least squares mean; Test type: Superiority or Other; p = 0.074, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = 0.34, 95% CI [-0.01 to 0.68], Standard Error of Mean 0.17 — Direction: nsNSAIDs minus celecoxib

11. Secondary Outcome: Modified Brief Pain Inventory Short Form (m-BPI-sf) - Pain Severity Question 4
Description: m-BPI-sf questionnaire assessed pain severity and pain interference with functional activities during the 24 hour follow-up period.
  Q4: Subject response to 'how much pain you have right now'. Scale: 0 = no pain to 10 = pain as bad as you can imagine
Time Frame: Days 2, 3 and 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 135 | 133
scores on a scale
  Day 2 (N = 134, 133) | 3.64 (2.05) | 4.23 (2.26)
  Day 3 (N =135, 131) | 2.58 (1.81) | 2.92 (1.78)
  Day 7 (N = 133, 125) | 1.14 (1.56) | 1.43 (1.55)
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Day 2 Least squares mean; Test type: Superiority or Other; p = 0.017, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = 0.58, 95% CI [0.11 to 1.05], Standard Error of Mean 0.24 — Direction: nsNSAIDs minus celecoxib
Statistical Analysis 2: Comparison: Celecoxib vs nsNSAIDs; Day 3 Least squares mean; Test type: Superiority or Other; p = 0.108, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = 0.34, 95% CI [-0.05 to 0.74], Standard Error of Mean 0.20 — Direction: nsNSAIDs minus celecoxib
Statistical Analysis 3: Comparison: Celecoxib vs nsNSAIDs; Day 7 Least squares mean; Test type: Superiority or Other; p = 0.117, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = 0.32, 95% CI [-0.01 to 0.66], Standard Error of Mean 0.17 — Direction: nsNSAIDs minus celecoxib

12. Secondary Outcome: Modified Brief Pain Inventory Short Form (m-BPI-sf) - Pain Severity Index
Description: m-BPI-sf questionnaire assessed pain severity and pain interference with functional activities during the 24 hour follow-up period.
  Pain severity index is the average of the pain severity questions 1 to 4. Scale: 0 = no pain to 10 = pain as bad as you can imagine
Time Frame: Days 2, 3 and 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 135 | 133
scores on a scale
  Day 2 (N = 134, 133) | 4.24 (1.66) | 4.48 (1.84)
  Day 3 (N = 135, 131) | 2.84 (1.61) | 3.26 (1.57)
  Day 7 (N = 133, 125) | 1.37 (1.47) | 1.68 (1.44)
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Day 2 Least squares mean; Test type: Superiority or Other; p = 0.229, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = 0.21, 95% CI [-0.17 to 0.60], Standard Error of Mean 0.20 — Direction: nsNSAIDs minus celecoxib
Statistical Analysis 2: Comparison: Celecoxib vs nsNSAIDs; Day 3 Least squares mean; Test type: Superiority or Other; p = 0.027, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = 0.40, 95% CI [0.05 to 0.75], Standard Error of Mean 0.18 — Direction: nsNSAIDs minus celecoxib
Statistical Analysis 3: Comparison: Celecoxib vs nsNSAIDs; Day 7 Least squares mean; Test type: Superiority or Other; p = 0.070, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = 0.33, 95% CI [0.01 to 0.65], Standard Error of Mean 0.16 — Direction: nsNSAIDs minus celecoxib

13. Secondary Outcome: Modified Brief Pain Inventory Short Form (m-BPI-sf) - Pain Interference Question 5A
Description: m-BPI-sf questionnaire assessed pain severity and pain interference with functional activities during the 24 hour follow-up period.
  Q5A: Subject response to 'how, during the past 24 hours, pain has interfered with your general activity. Scale: 0 = does not interfere to 10 = completely interferes
Time Frame: Days 2, 3 and 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 135 | 133
scores on a scale
  Day 2 (N = 134, 133) | 5.40 (2.52) | 5.37 (2.62)
  Day 3 (N = 135, 131) | 3.65 (2.64) | 4.07 (2.60)
  Day 7 (N = 133, 125) | 1.78 (2.13) | 1.90 (1.94)
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Day 2 Least squares mean; Test type: Superiority or Other; p = 0.954, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = -0.05, 95% CI [-0.64 to 0.53], Standard Error of Mean 0.30 — Direction: nsNSAIDs minus celecoxib
Statistical Analysis 2: Comparison: Celecoxib vs nsNSAIDs; Day 3 Least squares mean; Test type: Superiority or Other; p = 0.172, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = 0.41, 95% CI [-0.19 to 1.02], Standard Error of Mean 0.31 — Direction: nsNSAIDs minus celecoxib
Statistical Analysis 3: Comparison: Celecoxib vs nsNSAIDs; Day 7 Least squares mean; Test type: Superiority or Other; p = 0.541, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = 0.16, 95% CI [-0.30 to 0.62], Standard Error of Mean 0.24 — Direction: nsNSAIDs minus celecoxib

14. Secondary Outcome: Modified Brief Pain Inventory Short Form (m-BPI-sf) - Pain Interference Question 5B
Description: m-BPI-sf questionnaire assessed pain severity and pain interference with functional activities during the 24 hour follow-up period.
  Q5B: Subject response to 'how, during the past 24 hours, pain has interfered with your mood'. Scale: 0 = does not interfere to 10 = completely interferes
Time Frame: Days 2, 3 and 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 135 | 133
scores on a scale
  Day 2 (N = 134, 133) | 3.72 (2.95) | 3.64 (2.87)
  Day 3 (N = 135, 131) | 2.43 (2.41) | 2.38 (2.60)
  Day 7 (N = 133, 125) | 1.17 (2.06) | 1.26 (2.01)
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Day 2 Least squares mean; Test type: Superiority or Other; p = 0.924, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = -0.08, 95% CI [-0.75 to 0.58], Standard Error of Mean 0.34 — Direction: nsNSAIDs minus celecoxib
Statistical Analysis 2: Comparison: Celecoxib vs nsNSAIDs; Day 3 Least squares mean; Test type: Superiority or Other; p = 0.898, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = -0.06, 95% CI [-0.62 to 0.51], Standard Error of Mean 0.29 — Direction: nsNSAIDs minus celecoxib
Statistical Analysis 3: Comparison: Celecoxib vs nsNSAIDs; Day 7 Least squares mean; Test type: Superiority or Other; p = 0.655, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = 0.13, 95% CI [-0.33 to 0.60], Standard Error of Mean 0.24 — Direction: nsNSAIDs minus celecoxib

15. Secondary Outcome: Modified Brief Pain Inventory Short Form (m-BPI-sf) - Pain Interference Question 5C
Description: m-BPI-sf questionnaire assessed pain severity and pain interference with functional activities during the 24 hour follow-up period.
  Q5C: Subject response to 'how, during the past 24 hours, pain has interfered with your walking ability'. Scale: 0 = does not interfere to 10 = completely interferes
Time Frame: Days 2, 3 and 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 135 | 133
scores on a scale
  Day 2 (N = 134, 133) | 5.10 (2.76) | 5.11 (2.74)
  Day 3 (N = 135, 131) | 3.58 (2.62) | 3.69 (2.67)
  Day 7 (N = 133, 125) | 1.65 (2.19) | 1.62 (1.93)
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Day 2 Least squares mean; Test type: Superiority or Other; p = 0.929, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = 0.02, 95% CI [-0.59 to 0.62], Standard Error of Mean 0.31 — Direction: nsNSAIDs minus celecoxib
Statistical Analysis 2: Comparison: Celecoxib vs nsNSAIDs; Day 3 Least squares mean; Test type: Superiority or Other; p = 0.712, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = 0.11, 95% CI [-0.50 to 0.71], Standard Error of Mean 0.30 — Direction: nsNSAIDs minus celecoxib
Statistical Analysis 3: Comparison: Celecoxib vs nsNSAIDs; Day 7 Least squares mean; Test type: Superiority or Other; p = 0.993, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = 0.04, 95% CI [-0.44 to 0.51], Standard Error of Mean 0.24 — Direction: nsNSAIDs minus celecoxib

16. Secondary Outcome: Modified Brief Pain Inventory Short Form (m-BPI-sf) - Pain Interference Question 5D
Description: m-BPI-sf questionnaire assessed pain severity and pain interference with functional activities during the 24 hour follow-up period.
  Q5D: Subject response to 'how, during the past 24 hours, pain has interfered with your normal work (work outside the home and housework)'. Scale: 0 = does not interfere to 10 = completely interferes
Time Frame: Days 2, 3 and 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 135 | 133
scores on a scale
  Day 2 (N = 134, 133) | 5.29 (2.95) | 5.39 (2.76)
  Day 3 (N = 135, 131) | 4.04 (2.92) | 4.04 (2.88)
  Day 7 (N = 133, 125) | 1.84 (2.42) | 1.87 (2.11)
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Day 2 Least squares mean; Test type: Superiority or Other; p = 0.779, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = 0.11, 95% CI [-0.53 to 0.75], Standard Deviation 0.32 — Direction: nsNSAIDs minus celecoxib
Statistical Analysis 2: Comparison: Celecoxib vs nsNSAIDs; Day 3 Least squares mean; Test type: Superiority or Other; p = 0.972, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = -0.02, 95% CI [-0.69 to 0.65], Standard Error of Mean 0.34 — Direction: nsNSAIDs minus celecoxib
Statistical Analysis 3: Comparison: Celecoxib vs nsNSAIDs; Day 7 Least squares mean; Test type: Superiority or Other; p = 0.844, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = 0.07, 95% CI [-0.47 to 0.61], Standard Error of Mean 0.27 — Direction: nsNSAIDs minus celecoxib

17. Secondary Outcome: Modified Brief Pain Inventory Short Form (m-BPI-sf) - Pain Interference Question 5E
Description: m-BPI-sf questionnaire assessed pain severity and pain interference with functional activities during the 24 hour follow-up period.
  Q5E: Subject response to 'how, during the past 24 hours, pain has interfered with your relations with other people'. Scale: 0 = does not interfere to 10 = completely interferes
Time Frame: Days 2, 3 and 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 135 | 133
scores on a scale
  Day 2 (N = 134, 133) | 2.70 (2.78) | 2.67 (2.68)
  Day 3 (N = 135, 131) | 1.81 (2.26) | 1.69 (2.26)
  Day 7 (N = 133, 125) | 0.80 (1.70) | 0.78 (1.48)
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Day 2 Least squares mean; Test type: Superiority or Other; p = 0.944, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = -0.02, 95% CI [-0.63 to 0.60], Standard Error of Mean 0.31 — Direction: nsNSAIDs minus celecoxib
Statistical Analysis 2: Comparison: Celecoxib vs nsNSAIDs; Day 3 Least squares mean; Test type: Superiority or Other; p = 0.654, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = -0.12, 95% CI [-0.62 to 0.38], Standard Error of Mean 0.26 — Direction: nsNSAIDs minus celecoxib
Statistical Analysis 3: Comparison: Celecoxib vs nsNSAIDs; Day 7 Least squares mean; Test type: Superiority or Other; p = 0.952, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = 0.01, 95% CI [-0.36 to 0.39], Standard Error of Mean 0.19 — Direction: nsNSAIDs minus celecoxib

18. Secondary Outcome: Modified Brief Pain Inventory Short Form (m-BPI-sf) - Pain Interference Question 5F
Description: m-BPI-sf questionnaire assessed pain severity and pain interference with functional activities during the 24 hour follow-up period.
  Q5F: Subject response to 'how, during the past 24 hours, pain has interfered with your sleep'. Scale: 0 = does not interfere to 10 = completely interferes
Time Frame: Days 2, 3 and 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 135 | 133
scores on a scale
  Day 2 (N = 134, 133) | 2.97 (2.88) | 2.87 (2.64)
  Day 3 (N = 135, 131) | 1.90 (2.40) | 1.86 (2.28)
  Day 7 (N = 133, 125) | 0.68 (1.77) | 0.82 (1.61)
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Day 2 Least squares mean; Test type: Superiority or Other; p = 0.842, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = -0.03, 95% CI [-0.65 to 0.59], Standard Error of Mean 0.31 — Direction: nsNSAIDs minus celecoxib
Statistical Analysis 2: Comparison: Celecoxib vs nsNSAIDs; Day 3 Least squares mean; Test type: Superiority or Other; p = 0.828, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = -0.04, 95% CI [-0.57 to 0.49], Standard Error of Mean 0.27 — Direction: nsNSAIDs minus celecoxib
Statistical Analysis 3: Comparison: Celecoxib vs nsNSAIDs; Day 7 Least squares mean; Test type: Superiority or Other; p = 0.542, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = 0.12, 95% CI [-0.30 to 0.53], Standard Error of Mean 0.21 — Direction: nsNSAIDs minus celecoxib

19. Secondary Outcome: Modified Brief Pain Inventory Short Form (m-BPI-sf) - Pain Interference Question 5G
Description: m-BPI-sf questionnaire assessed pain severity and pain interference with functional activities during the 24 hour follow-up period.
  Q5G: Subject response to 'how, during the past 24 hours, pain has interfered with your enjoyment of life'. Scale: 0 = does not interfere to 10 = completely interferes
Time Frame: Days 2, 3 and 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 135 | 133
scores on a scale
  Day 2 (N = 134, 133) | 3.33 (3.17) | 2.99 (2.81)
  Day 3 (N = 135, 131) | 2.13 (2.69) | 2.06 (2.48)
  Day 7 (N = 133, 125) | 1.07 (1.98) | 1.10 (1.80)
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Day 2 Least squares mean; Test type: Superiority or Other; p = 0.404, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = -0.25, 95% CI [-0.92 to 0.42], Standard Error of Mean 0.34 — Direction: nsNSAIDs minus celecoxib
Statistical Analysis 2: Comparison: Celecoxib vs nsNSAIDs; Day 3 Least squares mean; Test type: Superiority or Other; p = 0.816, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = 0.02, 95% CI [-0.53 to 0.58], Standard Error of Mean 0.28 — Direction: nsNSAIDs minus celecoxib
Statistical Analysis 3: Comparison: Celecoxib vs nsNSAIDs; Day 7 Least squares mean; Test type: Superiority or Other; p = 0.837, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = 0.07, 95% CI [-0.37 to 0.52], Standard Error of Mean 0.23 — Direction: nsNSAIDs minus celecoxib

20. Secondary Outcome: Modified Brief Pain Inventory Short Form (m-BPI-sf) - Pain Interference Index
Description: m-BPI-sf questionnaire assessed pain severity and pain interference with functional activities during the 24 hour follow-up period.
  The pain interference index is the average of pain interference questions 5A to 5G. Scale: 0 = does not interfere to 10 = completely interferes
Time Frame: Days 2, 3 and 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 135 | 133
scores on a scale
  Day 2 (N = 134, 133) | 4.07 (2.34) | 4.01 (2.12)
  Day 3 (N = 135, 131) | 2.79 (2.15) | 2.83 (2.07)
  Day 7 (N = 133, 125) | 1.28 (1.81) | 1.33 (1.54)
Statistical Analysis 1: Comparison: Celecoxib vs nsNSAIDs; Day 2 Least squares mean; Test type: Superiority or Other; p = 0.887, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = -0.04, 95% CI [-0.54 to 0.45], Standard Error of Mean 0.25 — Direction: nsNSAIDs minus celecoxib
Statistical Analysis 2: Comparison: Celecoxib vs nsNSAIDs; Day 3 Least squares mean; Test type: Superiority or Other; p = 0.889, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = 0.04, 95% CI [-0.43 to 0.51], Standard Error of Mean 0.24 — Direction: nsNSAIDs minus celecoxib
Statistical Analysis 3: Comparison: Celecoxib vs nsNSAIDs; Day 7 Least squares mean; Test type: Superiority or Other; p = 0.738, ANCOVA — Overall p value; Terms for treatment and country; Mean Difference (Final Values) = 0.09, 95% CI [-0.30 to 0.47], Standard Error of Mean 0.20 — Direction: nsNSAIDs minus celecoxib

ADVERSE EVENTS:
Arm/Group | Celecoxib | nsNSAIDs
Serious Adverse Events (participants affected / at risk) | 0 | 2
Other Adverse Events (participants affected / at risk) | 13 | 17
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Celecoxib | nsNSAIDs
Dengue fever (Infections and infestations) | 0/141 | 1/137
Tendon rupture (Injury, poisoning and procedural complications) | 0/141 | 1/137
OTHER ADVERSE EVENTS (reported when occurring in more than 1.5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Celecoxib | nsNSAIDs
Abdominal pain upper (Gastrointestinal disorders) | 0/141 | 2/137
Diarrhoea (Gastrointestinal disorders) | 1/141 | 2/137
Dyspepsia (Gastrointestinal disorders) | 1/141 | 2/137
Gastritis (Gastrointestinal disorders) | 2/141 | 5/137
Hyperchlorhydria (Gastrointestinal disorders) | 1/141 | 3/137
Nausea (Gastrointestinal disorders) | 1/141 | 2/137
Headache (Nervous system disorders) | 3/141 | 0/137
Somnolence (Nervous system disorders) | 5/141 | 2/137

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.